CLINICAL TRIAL: NCT01371409
Title: Interhemispheric Contributions to Neuroplasticity and Motor Learning After Stroke
Brief Title: Interhemispheric Inhibitory Interactions
Acronym: InHIb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H09-00368; CIHR (Other Grant/Funding Number: 221612)
Record Dates: First submitted 2011-06-02; First posted 2011-06-10 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Stroke
Keywords: Stroke; TMS; Paired Pulse; EEG; Motor Learning
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active cTBS (Experimental)
  Interventions: Other: continuous theta burst stimulation
- Sham cTBS (Sham Comparator)
  Interventions: Other: continuous theta burst stimulation

INTERVENTIONS:
Other: continuous theta burst stimulation — 80% active motor threshold, 600 pulses
  Other Names: transcranial magnetic stimulation

SUMMARY:
After a stroke the excitability of the brain decreases on the stroke side and increases on the opposite, non-stroke side. These changes make use of the stroke-affected arm difficult and slow recovery. Rehabilitation exercises that increase arm use after stroke help increase brain excitability, but the net effect of this approach is low. New therapies are needed that restore more equal levels of brain excitability between the two sides. Brain stimulation is a noninvasive way to affect activity the excitability of brain cells. Pairing brain stimulation with exercises that require patients to learn new movements may help the brain to learn. Using stimulation that reduces activity in the side opposite to the stroke can increase activity on the stroke -affected side, through connections between the two brain hemispheres. The purpose of this study is to test if brain stimulation on the side opposite to the stroke, paired with arm movement exercises, can help patients learn new arm movements and improve arm function.

In this study people with stroke will receive brain stimulation over two different areas on the side of the brain opposite to the stroke: 1) those areas responsible for movement and 2) those responsible for sensation. These experiments will test both the short and long term effects of brain stimulation on patients' learning and arm function and will allow us to identify which area of the brain best improves learning and arm function. These experiments have the potential to improve the effectiveness of rehabilitation after stroke. The proposed study is among the first to test stimulation over the side of the brain opposite to the stroke damage and at multiple sites. This unique approach may help stimulate the development of new methods for stroke rehabilitation.

DETAILED DESCRIPTION:
The overall objective of this proposal is to examine the efficacy of new approaches to stroke recovery based on recent reports of interhemispheric contributions to neuroplastic change and motor skill learning. After stroke, cortical excitability is decreased in the ipsilesional and increased in the contralesional primary motor cortices (M1). Combined, these changes hamper hemiparetic arm use and impede functional recovery. Increasing hemiparetic arm use elevates the excitability of the ipsilesional cortex and improves function. Importantly, skilled motor practice raises cortical excitability to an even greater extent than merely increasing generalized use. However, the impact of increasing cortical excitability on recovery of function after stroke is limited, perhaps because the rate of change associated with both increasing use and learning new motor skills is low.

Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive method of brain stimulation. In humans, rTMS applied at high frequencies can increase cortical excitability; conversely, at low frequencies it can decrease cortical excitability. While rTMS in isolation can change cortical excitability after stroke its impact on neuroplastic change is small, likely reflecting a lack of consolidation in the absence of paired motor behaviour. Modulating the activity in a given neural network with brain stimulation prior to motor skill practice may in essence prime the system and enhance the neuroplastic effects associated with learning new motor skills. Yet to date, few studies have paired rTMS with practice of a novel motor task and assessed changes in motor function or behaviour.

Intuitively, it seems simplest to employ high frequency rTMS in the ipsilesional cortex to enhance cortical excitability. However, because of the difficulty of locating stimulation targets in the damaged hemisphere, low-frequency rTMS applied over the contralesional cortex may be the better approach. Though the direct effect of low-frequency rTMS in the human cortex is to suppress activity in the stimulated region it also indirectly enhances distant activity. Low-frequency rTMS over M1 increases cortical activity in the contralateral M1 homologue. We recently extended this finding to the primary sensory cortex (S1); demonstrating that low-frequency rTMS over left S1 increased excitability in (i.e., disinhibited) right S1. Therefore, suppressing the contralesional cortex to enhance ipsilesional cortical activity may facilitate a neural environment that is conducive for neuroplastic change.

Taken together these data suggest that inhibitory brain stimulation over the contralesional cortex, paired with skilled motor practice, may offer a new approach for stroke rehabilitation. To better understand whether this approach has merit, we propose to test two specific aims in separate experiments.

Specific Aim: To test the cumulative effects of repeated sessions that pair brain stimulation over M1c versus S1c with skilled motor practice in individuals with stroke.

We will assess hemiparetic arm motor and sensory function, motor performance/ motor skill acquisition (repeated sequence response times), cortical excitability, and neuroelectric activity in individuals with chronic sub-cortical stroke. Pre-brain stimulation measures will be compared with those obtained after 5 days of training paired with brain stimulation at a separate no-rTMS retention test to assess the cumulative effects of brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

* aged 40-75
* single, MCA territory stroke
* at least 6 months post stroke
* Fugl-Meyer (upper extremity) score of 15-55

Exclusion Criteria:

* absence of TMS motor evoked potential
* score <24 on the Montreal Cognitive Assessment
* history of seizure/epilepsy, head trauma, major psychiatric diagnosis
* aphasic (score <13 on Frenchay Aphasia Screen)
* contraindications to TMS/MRI

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Response Time | change from baseline to day 6
  Response time on a custom designed serial tracking program

SECONDARY OUTCOMES:
Wolf Motor | change from baseline to day 6
  standardized measure of upper limb function
Limb Position Matching | change from baseline to day 6
  Limb position matching using custom designed software
Intracortical Inhibition | change from baseline to day 6
  Intracortical Inhibition as measured by paired pulse transcranial magnetic stimulation
Movement Time | change from baseline to day 6
  movement time on custom designed serial tracking program
Movement Trajectory | change from baseline to day 6
  Movement trajectory on a custom designed serial tracking program
Intracortical facilitation | change from baseline to day 6
  Intracortical facilitation as measured by paired pulse transcranial magnetic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Lara A Boyd, PT, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided